CLINICAL TRIAL: NCT00262106
Title: An International Multi-centre, Randomised, Double-blind, Placebo-controlled Trial to Evaluate the Efficacy and Safety of 0.5% and 2% PRO 2000/5 Gels for the Prevention of Vaginally Acquired HIV Infection
Brief Title: Trial to Evaluate PRO 2000/5 Gels for the Prevention of Vaginally Acquired HIV Infection
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Endo Pharmaceuticals (Industry)
Collaborators: Medical Research Council (Other Government); Department for International Development, United Kingdom (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: MDP301; ISRCTN64716212
Record Dates: First submitted 2005-12-05; First posted 2005-12-06 (Estimated); Last update posted 2012-09-10 (Estimated); Status verified 2012-09

CONDITIONS: HIV Infections; Gonorrhea; Chlamydial Infections; Genital Herpes
Keywords: Administration, intravaginal; Anti-infective agents; Double blind method; Drug evaluation; Female; Gels; HIV infections/prevention and control; Microbicide; Naphthalenesulfonates/administration and dosage; Polymers/administration and dosage; Sexual behavior; Vaginal creams, foams and jellies; HIV Seronegativity; Genital Herpes Infections
MeSH Terms: conditions — HIV Infections; Gonorrhea; Chlamydia Infections; Herpes Genitalis; Sexual Behavior | interventions — naphthalenesulfonic acid, polymer with formaldehyde

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Placebo (Placebo Comparator): placebo
  Interventions: Drug: Placebo
- PRO 2000/5 Gel 0.5% (Active Comparator): PRO 2000/5 Gel 0.5%
  Interventions: Drug: PRO 2000/5

INTERVENTIONS:
Drug: PRO 2000/5 — Gel
  Arms: PRO 2000/5 Gel 0.5%
Drug: Placebo — Placebo
  Arms: Placebo

SUMMARY:
The objective of the study is to determine the efficacy and safety of 0.5% and 2% PRO 2000/5 gels compared to placebo in preventing vaginally acquired HIV infection.

DETAILED DESCRIPTION:
The HIV pandemic continues with an estimated 13,000 new infections each day, the vast majority of which are acquired through heterosexual intercourse. Although consistent and correct use of condoms by men remains the most effective form of protection from heterosexually acquired HIV, women are not always able to negotiate condom use. An effective prophylactic vaccine remains a key objective, but development is slow because of virus variability and difficulty in determining the immunological correlates of protection. Vaginal microbicides are being developed in response to the urgent need for an HIV prevention method that women can control. Licensed spermicides containing nonoxynol-9 (N-9), which has potent anti-HIV activity in vitro, were the first products to be investigated as potential microbicides. However, the association of N-9 and other products belonging to this class (surfactants) with genital epithelial disruption, histologically determined genital inflammation, and reduction in populations of vaginal lactobacilli led to concerns that their use could enhance the risk of HIV transmission. Early Phase 3 studies of N-9 products yielded conflicting results, but more recently, a multicenter randomized placebo-controlled trial of a low dose N-9 formulation demonstrated an increased incidence of HIV infection in the N-9 group compared to placebo. These findings have intensified efforts to develop agents with a more favorable toxicity profile. At least four of these have entered trials to assess effectiveness in preventing vaginally acquired HIV infection: Buffer Gel, Carraguard, cellulose sulfate and PRO 2000/5 Gel. Protocol MDP 301 describes a randomized placebo-controlled trial design to explore the safety and efficacy of two concentrations of PRO 2000/5 Gel.

Participant recruitment and follow-up is complete. Between October 2005 and August 2008, 9404 eligible, sexually active, HIV-uninfected women were enrolled at six or more sites in Africa. Up until February 2008, participants were randomly assigned to 0.5% or 2% PRO 2000/5 Gel treatment arms or a placebo gel arm. Following a recommendation by the Independent Data Monitoring Committee that the 2% PRO2000/5 Gel treatment arm should not continue as there was no more than a small chance of demonstrating benefit, participants enrolled after February 13, 2008 were randomly assigned to the 0.5% PRO 2000/5 gel treatment arm or placebo arm. Participants were instructed to apply a single dose of study gel 1 hour or less before every act of vaginal intercourse using a single-use pre-filled applicator. Participants also receive risk-reduction counseling and condoms, and STD testing. Most study participants were followed for 12 months. A cohort of sero-discordant couples enrolled in Uganda was followed for up to 24 months.

The primary efficacy outcome measure is acquisition of HIV infection at the 12 month time point. Secondary outcomes include measures of HIV infection at the 6, 9 and more than 12 month time points, infection by HSV-2, Neisseria gonorrhoeae, Chlamydia trachomatis, and adverse events.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 16 years and above at enrolment in Masaka and Mwanza, or aged 18 years and above at enrolment in the South African and Zambian sites
* Likely to be sexually active at entry and during follow-up
* Willing to undergo HIV testing at screening and approximately 12 weekly intervals, and additionally, if required, to determine HIV status
* HIV negative at screening according to the local HIV testing algorithm
* Willing to receive the HIV result before randomization
* Willing to use study gel as instructed
* Willing to undergo regular speculum examinations and genital infection screens
* Willing to have regular urine pregnancy tests
* Willing to receive health education about condoms
* Willing and able to give informed consent

Exclusion Criteria:

* Unable or unwilling to provide a reliable method of contact for the field team
* Likely to move permanently out of the area within the next year
* Likely to have sex more than 14 times a week on a regular basis during the course of follow-up
* Using spermicides regularly
* Pregnant or within 6 weeks postpartum at enrollment
* Has Grade 3 clinical or laboratory abnormalities which are considered by the clinician or the Trial Management Group to make enrollment inadvisable
* Requires referral for assessment of a clinically suspicious cervical lesion
* Treatment to the cervix, or to the womb through the cervix, within 30 days of enrolment
* Known latex allergy
* Participating, or has participated within 30 days of enrolment, in a clinical trial of an unlicensed product, microbicide, barrier method, or any other intervention likely to impact on the outcome of this trial
* Considered unlikely to be able to comply with the protocol

Min Age: 16 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 9404 (Actual)
Dates: Start 2005-10; Primary Completion 2008-08 (Actual); Study Completion 2009-09 (Actual)

PRIMARY OUTCOMES:
Acquisition of HIV infection before or at the 12 month time point, confirmed in a central laboratory, in participants confirmed to be HIV negative at enrollment | 12 months
Grade 3 (severe) or 4 (life-threatening) clinical or laboratory adverse event confirmed on examination or repeat testing, respectively | 12 months

SECONDARY OUTCOMES:
Acquisition of HIV infection before or at the 6, 9, or beyond 12 month time points, confirmed in a central laboratory, in participants confirmed to be HIV negative at enrollment | 6, 9 and 12 months
HSV-2 incidence rates by the 9 month time point in participants uninfected at enrollment. Although prevalence rates are high, 75% - 85% in some sites, data from feasibility studies indicate that incidence rates are also likely to be high | 9 months
HSV-2 incidence rates by the 12 month time point in participants uninfected at enrolment. Although prevalence rates are high, 75% - 85% in some sites, data from feasibility studies indicate that incidence rates are also likely to be high | 12 months
Cross-sectional prevalence of Neisseria gonorrhoeae at 24 weeks, determined by a positive nucleic acid amplification assay | 24 weeks/6 months
Cross-sectional prevalence of Chlamydia trachomatis at 24 weeks, determined by a positive nucleic acid amplification assay | 24 wks/6 months

CONTACTS AND LOCATIONS:
Overall Officials: Sheena McCormack, MBBS, MSc, FRCP, Principal Investigator — MRC Clinical Trials Unit
Locations (6):
- South Africa (3):
  - Reproductive Health and HIV Research Unit, Chris Hani Baragwanath Hospital, Bertsham
  - Africa Centre for Health and Population Studies, Mtubatuba
  - HIV Prevention Research Unit, Medical Research Council, Westville
- AMREF Lake Zone Programme, Mwanza, Tanzania
- MRC Programme on AIDS in Uganda, Uganda Virus Research Institute, Entebbe, Uganda
- MDP Zambia, Nakambala Sugar Estate, Mazabuka, Zambia

REFERENCES:
- [Background] Van Damme L, Wright A, Depraetere K, Rosenstein I, Vandersmissen V, Poulter L, McKinlay M, Van Dyck E, Weber J, Profy A, Laga M, Kitchen V. A phase I study of a novel potential intravaginal microbicide, PRO 2000, in healthy sexually inactive women. Sex Transm Infect. 2000 Apr;76(2):126-30. doi: 10.1136/sti.76.2.126. PMID 10858715
- [Background] Mayer KH, Karim SA, Kelly C, Maslankowski L, Rees H, Profy AT, Day J, Welch J, Rosenberg Z; HIV Prevention Trials Network (HPTN) 020 Protocol Team. Safety and tolerability of vaginal PRO 2000 gel in sexually active HIV-uninfected and abstinent HIV-infected women. AIDS. 2003 Feb 14;17(3):321-9. doi: 10.1097/00002030-200302140-00005. PMID 12556685
- [Background] Morrow K, Rosen R, Richter L, Emans A, Forbes A, Day J, Morar N, Maslankowski L, Profy AT, Kelly C, Abdool Karim SS, Mayer KH. The acceptability of an investigational vaginal microbicide, PRO 2000 Gel, among women in a phase I clinical trial. J Womens Health (Larchmt). 2003 Sep;12(7):655-66. doi: 10.1089/154099903322404302. PMID 14583106
- [Background] Tabet SR, Callahan MM, Mauck CK, Gai F, Coletti AS, Profy AT, Moench TR, Soto-Torres LE, Poindexter III AN, Frezieres RG, Walsh TL, Kelly CW, Richardson BA, Van Damme L, Celum CL. Safety and acceptability of penile application of 2 candidate topical microbicides: BufferGel and PRO 2000 Gel: 3 randomized trials in healthy low-risk men and HIV-positive men. J Acquir Immune Defic Syndr. 2003 Aug 1;33(4):476-83. doi: 10.1097/00126334-200308010-00008. PMID 12869836